CLINICAL TRIAL: NCT00003667
Title: Randomized Phase II Study of Vincristine, Doxorubicin, Cyclophosphamide and Dexrazoxane With and Without ImmTher for Newly Diagnosed High Risk Ewing's Sarcoma
Brief Title: Combination Chemotherapy and Biological Therapy in Treating Patients With High-Risk Ewing's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 98-074; CDR0000066764 (Registry Identifier: PDQ (Physician Data Query)); ENDOREX-MSKCC-98074; MDA-ID-97198; NCI-G98-1487
Record Dates: First submitted 1999-11-01; First posted 2004-06-24 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Sarcoma
Keywords: nonmetastatic childhood soft tissue sarcoma; metastatic childhood soft tissue sarcoma; extraosseous Ewing sarcoma/peripheral primitive neuroectodermal tumor; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Cyclophosphamide; Dexrazoxane; N-acetylglucosamine-N-acetylmuramyl-alanyl-isoglutaminyl-alanyl-glycerol dipalmitoyl; Doxorubicin; Vincristine; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: dexrazoxane hydrochloride
Drug: disaccharide tripeptide glycerol dipalmitoyl
Drug: doxorubicin hydrochloride
Drug: vincristine sulfate
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining chemotherapy with biological therapy may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of combination chemotherapy with or without biological therapy in treating patients who have newly diagnosed high-risk Ewing's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effects of dose intensive regimens of vincristine, doxorubicin, cyclophosphamide, and dexrazoxane with or without ImmTher (a muramyl dipeptide liposome) on the 2 year disease-free survival of patients with newly diagnosed high risk Ewing's sarcoma. II. Evaluate the feasibility and determine the toxicity of administering weekly ImmTher for 1 year to these patients. III. Determine which therapy is worthy of further evaluation.

OUTLINE: This is a randomized study. Patients are stratified according to the presence of bony metastases at diagnosis. Patients are randomized to one of two treatment arms. All patients receive dexrazoxane IV followed 30 minutes later by doxorubicin IV over 30 minutes on day 1, vincristine IV on day 1, and cyclophosphamide IV over 6 hours on days 1 and 2. Treatment is repeated every 3 weeks for 3-6 courses in the absence of disease progression or unacceptable toxicity. Patients are evaluated after course 3 and undergo surgery and/or radiation therapy. The next 3 courses of chemotherapy are administered after recovery from surgery/radiation therapy. Within 1 month after completion of all chemotherapy courses, patients randomized to arm I receive ImmTher IV over 60 minutes weekly for 1 year. Patients randomized to arm II receive no further therapy. Patients are followed every 6 weeks for 2 years.

PROJECTED ACCRUAL: A total of 105 patients will be accrued for this study within approximately 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven high risk Ewing's family of tumors: Ewing's sarcoma of bone Extraosseous Ewing's sarcoma Peripheral neuroepithelioma Must have one of the following characteristics: Metastatic disease at diagnosis Primary tumor of the humerus, femur, or trunk Bulky (greater than 8 cm) tumor Elevated LDH prior to biopsy (at least 900 IU/mL)

PATIENT CHARACTERISTICS: Age: 3 to 60 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Granulocyte count at least 500/mm3 Platelet count at least 75,000/mm3 Hemoglobin at least 8 g/dL (transfusion allowed) Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT or SGPT no greater than 3 times normal Renal: BUN less than 30 mg/dL Creatinine no greater than 1.5 times normal for age OR Creatinine clearance at least 70 mL/min Cardiovascular: Ejection fraction at least 50% OR Fractional shortening at least 29% Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-09; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Meyers, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas